CLINICAL TRIAL: NCT07203456
Title: Testing Educational Modalities for Temporomandibular Disorders Curriculum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: #IRB-24-0018
Record Dates: First submitted 2025-06-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Confidence; Diagnostic Ability

STUDY DESIGN:
Intervention Model Description: Educational intervention with virtual patient learning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical exposure to patients with TMD (Active Comparator): Participants will be exposed to clinical patients with TMD
  Interventions: Other: Clinical exposure to patients with TMD
- Clinical exposure to patients with TMD and virtual patient based learning (VPBL) (Active Comparator): Participants will be exposed to clinical patients with TMD and to the corresponding virtual patient with the same TMD diagnosis featured on the VPBL
  Interventions: Other: Clinical exposure to TMD + VPBL
- Virtual Patient Based Learning (VPBL) (Experimental): Participants will be exposed to review virtual patients featured on the VPBL
  Interventions: Other: Virtual Patient Based Learning (VPBL)

INTERVENTIONS:
Other: Virtual Patient Based Learning (VPBL) — A digital platform featuring 20 virtual patients has been built to increase predoctoral student clinical exposure to patients with TMD signs and symptoms
  Arms: Virtual Patient Based Learning (VPBL)
Other: Clinical exposure to patients with TMD — Participants in this arm will be exposed to patients with TMD signs and symptoms, to the history taking, interview, clinical examination, diagnostic process, and treatment plan under the supervision of an orofacial pain specialist
  Arms: Clinical exposure to patients with TMD
Other: Clinical exposure to TMD + VPBL — Participants will be exposed to patients with TMD signs and symptoms (including history taking, interview, clinical exam, diagnostic process, and treatment plan) under the supervision of an orofacial pain specialist, and then will be exposed to the corresponding TMD patient on the VPBL, featuring virtual patients with TMD
  Arms: Clinical exposure to patients with TMD and virtual patient based learning (VPBL)

SUMMARY:
This study is done to assess the change in confidence level, knowledge, and diagnostic ability in TMD-related aspects through the exposure to a Virtual Patient-Based Learning (VPBL) platform featuring temporomandibular disorder (TMD) cases among 3rd and 4th year predoctoral dental students at a larger predoctoral school.

ELIGIBILITY:
Inclusion Criteria:

* Third or Fourth year dental students at the College of Dental Medicine at Midwestern University (Illinois)

Exclusion Criteria:

* Dental students not enrolled at the third and/or fourth year of the College of Dental Medicine at Midwestern University (Illinois)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Self-perceived Confidence Level | Immediately after the educational intervention
  Change in confidence level between baseline and after the educational intervention. The self-perceived confidence level will be measured with a 12-item confidence level scale (previously developed and validated by the research group), where answer options range from 0 to 10 on a numerical rating scale (with 0 = "not confident at all" and 10 = "extremely confident"). The 12 items refer to TMD-related skills, including but not limited to providing a treatment plan for patients with TMD, screening of TMD patients, education on the TMD condition, performing diagnostic injections, referring to healthcare providers, among others.

SECONDARY OUTCOMES:
Diagnostic ability in diagnosing TMD cases | Immediately after the educational intervention
  Change in diagnostic ability in TMD. The diagnostic ability in TMD will be assessed by providing case scenarios featuring signs and symptoms of various TMD conditions. The user will be asked to indicate the TMD diagnosis of the described case. Diagnostic ability will be evaluated based on the accuracy of identifying the correct TMD condition based on the Diagnostic Criteria for TMD (DC/TMD). Answers will be given a score of 1 in case of accurate diagnosis and 0 in case of inaccurate diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No